CLINICAL TRIAL: NCT04692961
Title: Change in the Lower Leg Muscle Stiffness Following Peroneal Artery-based Flap: An Elastography Ultrasonographic Study
Brief Title: Change in the Lower Leg Muscle Stiffness Following Peroneal Artery-based Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202009077RIND
Record Dates: First submitted 2020-12-23; First posted 2021-01-05 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2023-02

CONDITIONS: Donor Site Complication; Muscle; Ischemic
Keywords: Elastography; Donor site morbidity
MeSH Terms: conditions — Ischemia | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients after free flap harvested (Experimental): Patients receiving peroneal artery-based free flap harvest
  Interventions: Device: Elastography

INTERVENTIONS:
Device: Elastography — Use elastography to evaluate the stiffness of lower leg muscle after peroneal artery-based free flap harvested

SUMMARY:
In the field of reconstructive microsurgery, donor site morbidity after free flap harvest is one of the key factors to consider when choosing among different options of free flap. Peroneal artery-based free flap, such as fibula flap or peroneal flap, is one of the popular options of free flap. There are a plenty of literature using a variety of modalities to evaluate the donor site morbidity after free fibula harvest, such as gait analysis. Elastography has been used to evaluate the stiffness change of soft tissue, such as skeletal muscle, or liver. The purpose of this study is to use elastography to evaluate the stiffness of lower leg muscle after peroneal artery-based free flap harvest.

DETAILED DESCRIPTION:
A total of twenty-three patients will be recruited at National Taiwan University Hospital Yunlin Branch. All of them will receive fibula flap or peroneal flap harvest operations. At the time points of pre-operation, 1-month post-operation, 3-month post-operation, and 6-month post-operation, the muscles of both legs of each patient will be evaluated by elastography, and the function of both legs will be evaluated by American Orthopedic Foot and Ankle Score (AOFAS). Paired t-test will be used to compare the results of each evaluations.

ELIGIBILITY:
Inclusion Criteria:

* No previous major operations over both legs
* Able to walk freely during daily life
* Going to receive peroneal artery-based free flap harvested from one leg

Exclusion Criteria:

* Previous major operations over either leg
* Unable to walk freely during daily life

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Lower Leg Muscle stiffness | 6 months
  Lower leg muscle stiffness after peroneal artery-based flap harvested; Name of measurement: elastic modulus; Unit: kPa

SECONDARY OUTCOMES:
American Orthopedic Foot and Ankle (AOFAS) scale | 6 months
  AOFAS scale change after peroneal artery-based flap harvested, highest score:100, lowest score: 0; A higher score means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Sheng Lin, MD, MPH, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Yunlin Branch, Douliu, Yunlin County, Taiwan

IPD SHARING:
Plan to Share IPD: No